CLINICAL TRIAL: NCT01354236
Title: Psychosocial Risk- and Protective Factors of Secondary School Dropout in Luxembourg: an Exploratory Case-control Study
Brief Title: Mental Health Related to School Dropout in Luxembourg
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Public Research Centre Health, Luxembourg (Other)
Collaborators: Fonds National de la Recherche Scientifique (Other); Université de Liège (Other); Hôpital du Kirchberg (Unknown); Ministère de l'Education nationale et de la Formation professionnelle (Unknown)
Responsible Party: Pascale Esch, Public Research Centre Health, Luxembourg
Other Study IDs: AFR-CESP-20100403
Record Dates: First submitted 2011-05-11; First posted 2011-05-16 (Estimated); Last update posted 2011-05-16 (Estimated); Status verified 2011-05

CONDITIONS: Anxiety Disorders; Mood Disorders; Eating Disorders; Substance-related Disorders; Impulse Control Disorders; Psychotic Disorders; Antisocial Personality Disorder
MeSH Terms: conditions — Anxiety Disorders; Mood Disorders; Feeding and Eating Disorders; Substance-Related Disorders; Disruptive, Impulse Control, and Conduct Disorders; Psychotic Disorders; Antisocial Personality Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- School dropouts: Students who quit school without graduation
- Controls: Normally enrolled students matched for age, gender, school and educational level

SUMMARY:
This study aims to investigate psychosocial risk- and protective factors such as psychiatric disorder, socio-economic background and family functioning among school dropouts and to compare the findings with those by a matched control group of regularly enrolled students.

DETAILED DESCRIPTION:
In Luxembourg, the national authorities had to face school dropout rates of more than 15%. As a result, they introduced accompanying and preventive measures to reduce linguistic and cultural risk factors that may impede educational engagement and vocational decisions. Since 2006, the dropout rate has overall declined. However the proportion of early school leavers who remain without any specific occupation is still alarming.

This study aims to identify psychosocial risk - and protective factors of secondary school dropout in order to deliver solid insight on how to tailor early detection and intervention programs.

In the light of prior findings, the investigators hypothesize that school dropouts have significantly more mental health problems than their peers who go to school. They are also more likely to report a poor socio-economic background, negative school experiences and difficulties in family functioning.

To test those hypotheses, the investigators will have an exploratory case control study.Recruitment of cases will be prospective, from an exhaustive population of dropouts and recruitment of matched controls will be done by random sampling. Data will be collected using self-report questionnaires on mental health, family life and problematic internet use as well as a structured clinical interview to consider psychiatric diagnosis according to the criteria of DSM IV.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in a public secondary school in Luxembourg
* Cases have to be reported as "school dropouts" in the electronic records of the ministry for education
* Informed consent obtained and signed by the adolescent and his/her legal guardian if the participant hasn't reached full age
* Understand German or French, which are the two languages of testing
* Resident in Luxembourg

Exclusion Criteria:

* Acute hospitalization or arrest

Ages: 16 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Cases: The ministry for education retrieves a monthly record of students classified as "school dropouts", who will be individually invited to participate in the study.
  Controls: Normally enrolled students who are matched for age, gender, school and educational grade. Their recruitment will be subsequent to the participation of cases.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2011-01

PRIMARY OUTCOMES:
Prevalence and type of psychiatric disorders | 1.5 years
  Odds ratios of psychiatric disorders between cases and controls

SECONDARY OUTCOMES:
Family variables (task fulfillment,role performance, communication, affective expression, connectedness, control behaviour, values and standards) | 1.5 years
  Odds ratios of family variables as predictors of interest and school dropout. As associations between the primary outcome measure and school dropout may vary with family variables, interactions between family variables and classes of mental disorders will be analyzed.
Socio-economic background (low, medium, high) | 1.5 years
  Odds ratios of socio-economic background as predictor of interest and school dropout. As associations between psychiatric disorders and school dropout may vary with socio-economic background, interactions between socio-economic background and classes of mental disorders will be analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Lise Lair, Study Director — Public Research Centre Health, Luxembourg; Pascale Esch, Principal Investigator — Public Research Centre Health, Luxembourg
Locations (1):
- Public Research Centre Health, Luxembourg, Strassen, Luxembourg

REFERENCES:
- [Derived] Esch P, Bocquet V, Pull C, Couffignal S, Graas M, Lair ML, Lehnert T, Fond-Harmant L, Ansseau M. Psychosocial risk and protective factors of secondary school dropout in Luxembourg: the protocol of an exploratory case-control study. BMC Public Health. 2011 Jul 13;11:555. doi: 10.1186/1471-2458-11-555. PMID 21752239